CLINICAL TRIAL: NCT06204770
Title: a Prospective, Single-arm, Symptom-based Score, to Evaluate the Tolerance of Extensive Hydrolyzed Whey Protein Milk Intervention Among Infant With Mild to Moderate CMPA
Brief Title: Tolerance of Extensive Hydrolyzed Whey Protein Milk Among Infant With Mild to Moderate CMPA
Acronym: PEACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was discontinued following the death of the Principal investigator
Sponsor: Danone Specialized Nutrition Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 180923
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Mild to Moderate Cows' Milk Protein Allergy

STUDY DESIGN:
Intervention Model Description: Participants will be asked to use NR Pepti as part their management of mild to moderate Cow's milk protein allergy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- groups of infants with CMPA (Experimental): Administered treatment for 4 weeks during intervention period.
  Interventions: Other: extensive hydrolyzed protein formula

INTERVENTIONS:
Other: extensive hydrolyzed protein formula — NR Pepti is infant formula for special medical purposes based on extensive hydrolyzed whey protein for infants aged 0-12 months. This milk is intended for cow's milk protein allergy. This product is lactose free with medium chain triglycerides (MCT)

SUMMARY:
The goal of this clinical trial is to evaluate the tolerance, safety and efficacy of Nutribaby Royal Pepti Junior (NR Pepti) among infants with mild to moderate Cow's Milk Protein Allergy (CMPA).

The main questions it aims to answer are:

1. Is NR Pepti tolerable among infants with mild to moderate CMPA?
2. Is NR Pepti safe and effective among infants with mild to moderate CMPA?

Participants will be asked to use NR Pepti as part their management of mild to moderate CMPA

DETAILED DESCRIPTION:
This study will be carried out by a principal investigator and co-investigators, all of whom will collaborate with doctors from Indonesian Pediatric Society (IDAI) in the Jakarta, Bogor, Depok, Tangerang and Bekasi (Jabodetabek) area. The following is the flow of subject recruitment:

1. Investigators will make direct contact with their patients and also recruit subjects through referral from IDAI pediatricians in the Jabodetabek area who have potential eligible patients for this study.
2. The media to be used in the recruitment are leaflets which firstly will be reviewed by the Ethics Committee. The leaflet will summarize information regarding the study and the referral procedures.
3. If the pediatrician has a subject that meets the eligibility criteria, they may reach the Principal Investigator (PI) or Study Team.
4. The Study Team will arrange discussion between pediatricians and the study team. The investigators will then carry out a brief assessment on the subject's inclusion and exclusion criteria.
5. If declared feasible and IDAI's pediatricians agree to refer their subject(s), the study team will coordinate with the pediatricians about their status in the study, and will coordinate with the subject to assign them to one of the listed sites run by investigators.
6. After the subject is completely transferred to the study site, the investigator will perform an informed consent process and continue by assessing the subject's inclusion and exclusion criteria on site.
7. If the assessment passed, the study team can start to intervene on the subject according to the provisions of the protocol.
8. During the intervention period, the study team will be assisted by Study Coordinator (SC) in maintaining the availability of milk investigational products for the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients (3-11 months) that are diagnosed with mild and moderate CMPA by HCPSs (Health Care Professional) having ≥ 1 symptoms such as:

   * Gastrointestinal: Frequent regurgitation, Vomiting, Diarrhea, Constipation, Blood in stool without failure to thrive
   * Dermatological: Atopic dermatitis, Swelling of lips or eyelids, Urticaria unrelated to acute infections, drug intake, or other causes
   * Respiratory: Runny nose, Recurrent otitis media, Chronic cough, Broncho-constriction unrelated to infection
   * General: Persistent distress, Colic (≥ 3 h/day wailing/irritable) over a period of > 3 weeks CMPA patients who have another food allergy are still allowed to participate in this study.
2. Subjects consumed only formula or mixed feeding (breast milk and formula milk, with maximum two times of breastfeeding in a day). Subject consuming weaning or complementary food is still allowed.
3. Mothers with mix-fed children willing to eliminate consuming any cow's milk product during the mix-fed period to avoid allergy onset due to breast milk.
4. Subject willing to stop any other formula while participating in this study
5. Subject willing to adhere to the investigator's prescription for daily IP consumption during the study.
6. Every patient that has been diagnosed with symptom-based CMPA must also have a record of being treated by consultant's ≥ 2 times for the past 2 weeks before screening (the 2nd consultation could also be on the screening visit).
7. Every patient needs to have at least 1 diagnosis result to confirm symptom-based CMPA. (Previous diagnosis methods could be used if available. If previous result is not available, HCP will perform one of the method mention in the protocol, the chosen diagnosis method is given to the HCP to be determined).
8. At the screening visit, the patient's SBS score must be minimum 1.

Exclusion Criteria:

1. Pediatric patients who have other immunologic disorders history.
2. Pediatric patients with congenital metabolic disorders, anatomic abnormalities, celiac disease, pancreatic insufficiency (cystic fibrosis), lactose intolerance, non-allergic gastro esophageal reflux disease, malignancy, and infection (Differential Diagnosis).

Ages: 3 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
evaluate tolerance of NR Pepti among infants with mild to moderate CMPA. | during the study period 28 days
  NR Pepti is determined to have tolerance if, during the 28 days of formula ingestion, there is no new symptom or developing allergic reaction as assessed by Symptom-Based Score Questionnaire that was developed by Vanderplas, et. al (2013) in 90% of the population compared to baseline.
  New symptom is described as CMPA symptoms that appear in the SBS questionnaire during the study while not being appeared in the baseline.
  Developing allergy reaction is describe as increase of existing CMPA symptom grade as assessed using SBS questionnaire during the study compared to the baseline

SECONDARY OUTCOMES:
evaluate the safety of NR Pepti among infants with mild to moderate CMPA. | during the study period 28 days
  Safety is measured by the number of participants with treatment-related adverse event as assessed by CTCAE v.5.0
evaluate the efficacy of NR Pepti among infants with mild to moderate CMPA. | during the study period 28 days
  Efficacy is measured by Symptom-Based Score (SBS) Questionnaire that was developed by Vanderplas, et. al (2013), with range score varies from 0 to 33.
  NR Pepti is determined to have efficacy if, during the 28 days of formula ingestion, there is ≥50% decrease of SBS score in all of enrolled subjects compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nia Kurniati, PhD, Principal Investigator — Pediatric Department, Faculty of Medicine, Universitas Indonesia
Locations (5):
- Indonesia (5):
  - Prof. Dr. dr. Zakiudin Munasir, Sp.A (K)'s private clinic, Tangerang, Banten
  - Siloam Hospital Lippo Vilage, Tangerang, Banten
  - dr. Martani Widjajanti Sukarlan, Sp.A (K)'s private clinic, Jakarta, DKI Jakarta
  - RSUPN Dr. Cipto Mangunkusumo Kencana and Kiara, Jakarta, DKI Jakarta
  - Hermina Hospital Depok, Depok, West Java

IPD SHARING:
Plan to Share IPD: No
will be discussed with principal investigator